CLINICAL TRIAL: NCT05633537
Title: Clinical and Radiographic Evaluation of Zinc Oxide-Ozonated Oil as a New Root Canal Filling Material for Primary Molars
Brief Title: Clinical & Radiographic Evaluation of Zinc Oxide-Ozonated Oil as a New Primary Root Canal Filling
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Shaimaa Shaban Mohamed El-desouky, Lecturer of Pediatric dentistry, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: #R- PED-1-21-2
Record Dates: First submitted 2022-11-21; First posted 2022-12-01 (Actual); Last update posted 2023-12-07 (Actual); Status verified 2023-12

CONDITIONS: Pulp Disease, Dental; Obturation; Root Canal Infection
Keywords: pulpectomy; Ozonated Olive Oil; zinc oxide eugenol; primary molars
MeSH Terms: conditions — Dental Pulp Diseases; Bites and Stings

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- group 1: zinc oxide-ozonated olive oil (Experimental): Group I: 30 primary molars were filled with fresh mix of zinc oxide powder with ozonated olive oil
  A single-visit pulpectomy procedure was performed . Standardized preoperative periapical radiograph was obtained to assess tooth condition & proper selection. Teeth were anesthetized & Rubber dam isolation was done, then all caries was removed & access opening was gained. Working length was determined by apex locator. All canals were prepared using Kidzo file system in a lateral brushing motion with an Endo-Mate DT endodontic motor at 350 RPM and 2.5 N/cm torque. EDTA gel 17% will be used before instrumentation & irrigation was done with normal saline. Dryness with paper points size 30 . placement of the root canal filling material (zinc oxide-ozonated olive oil) was applied . Intermediate restorative material was placed, then tooth was restored with stainless-steel crown
  Interventions: Procedure: pulpectomy procedure and the clinical evaluation; Radiation: radiographic evaluation
- group 2: zinc oxide- olive oil (Experimental): Group 2: 30 primary molars were filled with fresh mix of zinc oxide powder with olive oil
  A single-visit pulpectomy procedure was performed . Standardized preoperative periapical radiograph was obtained to assess tooth condition & proper selection. Teeth were anesthetized & Rubber dam isolation was done, then all caries was removed & access opening was gained. Working length was determined by apex locator. All canals were prepared using Kidzo file system in a lateral brushing motion with an Endo-Mate DT endodontic motor at 350 RPM and 2.5 N/cm torque. EDTA gel 17% will be used before instrumentation & irrigation was done with normal saline. Dryness with paper points size 30 . placement of the root canal filling material (zinc oxide- olive oil) was applied . Intermediate restorative material was placed, then tooth was restored with stainless-steel crown
  Interventions: Procedure: pulpectomy procedure and the clinical evaluation; Radiation: radiographic evaluation
- group 3:zinc oxide- eugenol (Active Comparator): Group 3: 30 primary molars were filled with zinc oxide- eugenol
  A single-visit pulpectomy procedure was performed . Standardized preoperative periapical radiograph was obtained to assess tooth condition & proper selection. Teeth were anesthetized & Rubber dam isolation was done, then all caries was removed & access opening was gained. Working length was determined by apex locator. All canals were prepared using Kidzo file system in a lateral brushing motion with an Endo-Mate DT endodontic motor at 350 RPM and 2.5 N/cm torque. EDTA gel 17% will be used before instrumentation & irrigation was done with normal saline. Dryness with paper points size 30 . placement of the root canal filling material (zinc oxide- eugenol) was applied . Intermediate restorative material was placed, then tooth was restored with stainless-steel crown
  Interventions: Procedure: pulpectomy procedure and the clinical evaluation; Radiation: radiographic evaluation

INTERVENTIONS:
Procedure: pulpectomy procedure and the clinical evaluation — in this study, pulpectomy procedure was performed in a single visit and the root canals were filled with different obturating materials. The clinical follow up evaluation was carried out after three, six and twelve months after pulpectomy procedures. The teeth were clinically evaluated each follow up visit for the following clinical features: absence of spontaneous pain, no tenderness with percussion, no abnormal mobility and absence of swelling & sinus or fistula. If the tooth exhibited any one of above clinical features, the pulpectomy was considered to be a failure (F); otherwise, it was regarded as clinical success (S).
  Other Names: clinical evaluation of root canal treatment of primary molars
Radiation: radiographic evaluation — Radiographic evaluation was performed immediately after teeth restoration (base line radiograph), then after three, six and twelve months. The parallel periapical technique was performed using the rinn (XCP) periapical film holder and a long cone which was mounted to the x-ray tube. The criteria for radiographic success were no evidence of extensive pathologic root resorption, reduction or no change in pre-operative pathologic inter-radicular radiolucency and no evidence of new postoperative pathologic radiolucency.

SUMMARY:
Preserving primary teeth is essential for many aspects such as the child's growth and development, esthetic, functional, psychological, and dental arch integrity aspects. a randomized blinded controlled clinical trial aimed to evaluate the clinical and radiographic success of Zinc Oxide-Ozonated Olive Oil as root canal filling materials for primary molars compared to Zinc Oxide-Olive Oil & Zinc Oxide-eugenol. 90 primary molars of 30 children aged between 4-8 years with pulpally involved primary molars, are equally divided into 3 groups which treated with Zinc Oxide-Ozonated Olive Oil , zinc oxide -olive oil and zinc oxide eugenol as obturation materials following pulpectomy procedure. The subjects were followed up clinically and radiographically at 3, 6 and 12 months.

DETAILED DESCRIPTION:
Pulpectomy for primary teeth involves root canal preparation followed by obturation with a resorbable material. Zinc oxide eugenol (ZOE) is the most widely used obturating material. The main ZOE disadvantages are the difference in rate of resorption compared to the root, and limited antimicrobial activity. ZOE is formed when crude eugenol is mixed with zinc oxide. the set material easily hydrolyzes, resulting in free eugenol release which can be harmful to human soft tissues; this motivated the search for a new eugenol substitute to be combined with zinc oxide. Olive oil is a vegetable oil that comprises antioxidants, carotenoids, oleuropein, and oleocanthal, a phenolic component that significantly contributes to its antibacterial and anti-inflammatory properties. ozone in the form of ozonated olive oil, have the ability to produce nascent oxygen deep into the treated area without triggering irritation so, improved rheological characteristics, increased intracellular ATP, stimulated cellular metabolism, and expression of cytokines related to healing, particularly Transforming Growth Factor.

ELIGIBILITY:
Inclusion Criteria:

* Healthy & cooperative child
* history of spontaneous pain
* Percussion sensitivity
* presence of inter-radicular or periapical radiolucency
* No internal root resorption
* External root resorption limited to apical third and with at least two-thirds root intact.

Exclusion Criteria:

* Uncooperativeness of child and/or parents
* Unrestorable tooth
* Presence of calcific metamorphosis inside root canals
* Tooth with evidence of extensive internal/external pathological root resorption.

Ages: 4 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 90 (Actual)
Dates: Start 2021-07-04 (Actual); Primary Completion 2023-03-01 (Actual); Study Completion 2023-05-29 (Actual)

PRIMARY OUTCOMES:
clinical success of primary molar pulpectomy after using new root canal filling materials (Zinc Oxide-Ozonated olive Oil , Zinc Oxide- olive Oil) compared to the widely used material (zinc oxide material) | 12 months
  by assessing the presence or absence of spontaneous pain, presence or absence of tenderness with percussion, presence or absence of abnormal mobility and presence or absence of swelling and/or fistula during the follow-up intervals ( three, six and twelve months )
radiographic success of primary molar pulpectomy after using new root canal filling materials (Zinc Oxide-Ozonated olive Oil , Zinc Oxide- olive Oil) compared to the widely used material (zinc oxide material) | 12 months
  by assessing the presence or absence of extensive pathologic root resorption, reduction or no change in pre-operative pathologic inter-radicular radiolucency and presence or absence of new postoperative pathologic radiolucency. the assessment is done using periapical radiographs at three, six and twelve months after pulpectomy procedure.

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta University, Tanta, Gharbia Governorate, Egypt

REFERENCES:
- [Background] Barja-Fidalgo F, Moutinho-Ribeiro M, Oliveira MA, de Oliveira BH. A systematic review of root canal filling materials for deciduous teeth: is there an alternative for zinc oxide-eugenol? ISRN Dent. 2011;2011:367318. doi: 10.5402/2011/367318. Epub 2010 Oct 17. PMID 21991471
- [Background] Chandra SP, Chandrasekhar R, Uloopi KS, Vinay C, Kumar NM. Success of root fillings with zinc oxide-ozonated oil in primary molars: preliminary results. Eur Arch Paediatr Dent. 2014 Jun;15(3):191-5. doi: 10.1007/s40368-013-0094-8. Epub 2013 Nov 6. PMID 24197970
- [Background] Sarrami N, Pemberton MN, Thornhill MH, Theaker ED. Adverse reactions associated with the use of eugenol in dentistry. Br Dent J. 2002 Sep 14;193(5):257-9. doi: 10.1038/sj.bdj.4801539. PMID 12353045
- [Background] Ulusoy OI, Ekici MAG, Alacam T, Bari E, Ulusoy C. Virgin Olive Oil, Soybean Oil, and Hank's Balanced Salt Solution Used as Storage Media on Periodontal Ligament Cell Viability. Pediatr Dent. 2019 Nov 15;41(6):485-488. PMID 31882036
- [Background] Saini R. Ozone therapy in dentistry: A strategic review. J Nat Sci Biol Med. 2011 Jul;2(2):151-3. doi: 10.4103/0976-9668.92318. PMID 22346227